CLINICAL TRIAL: NCT00505635
Title: Biochemotherapy With Temozolomide, Velban, Cisplatin, Interleukin-2, Interferon-alpha and Thalidomide for Metastatic Melanoma With Optional Intrathecal Interleukin-2 Treatment
Brief Title: Biochemotherapy With Temozolomide for Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM03-0218
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Results first posted 2012-04-18 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Melanoma
Keywords: advanced stage IV melanoma; unresectable stage III melanoma; Melanoma; Temozolomide; Velban; Vinblastine; Cisplatin; Interleukin-2; Intron-A; Interferon Alpha-2b; Thalidomide; Thalomid; Temodar; Proleukin
MeSH Terms: conditions — Melanoma | interventions — Temozolomide; Vinblastine; Cisplatin; Interleukin-2; aldesleukin; Introns; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biochemotherapy with Temozolomide (Experimental): Temozolomide 250 mg/m^2 every 4 hours Day 1; Biochemotherapy of Velban 1.5 mg/m^2 intravenous (IV) Days 1-4; Cisplatin 20 mg/m^2 IV Days 1-4; + Interleukin-2 9 MIU/m^2 IV over 24 Hours for 4 Doses Days 1-4; Intron-A 5 mu/m^2 subcutaneously daily Days 1-5; + Oral Thalidomide 400 mg daily.
  Interventions: Drug: Temozolomide; Drug: Velban; Drug: Cisplatin; Drug: Interleukin-2; Drug: Intron-A; Drug: Thalidomide

INTERVENTIONS:
Drug: Temozolomide — 250 mg/m^2 By Mouth Every 4 Hours x 3 Doses On Day 1
  Other Names: Temodar
Drug: Velban — 1.5 mg/m^2 By Vein Over 15-30 Minutes On Days 1-4
  Other Names: Vinblastine
Drug: Cisplatin — 20 mg/m^2 By Vein Over 45-120 Minutes On Days 1-4
  Other Names: Platinol-AQ; Platinol; CDDP
Drug: Interleukin-2 — 9 MIU/m^2 By Vein Over 24 Hours x 4 Doses On Days 1-4
  Other Names: Proleukin; IL-2
Drug: Intron-A — 5 mu/m^2 Subcutaneously (Under the skin) Daily On Days 1-5
  Other Names: Interferon Alpha-2b
Drug: Thalidomide — 400 mg By Mouth Daily
  Other Names: Thalomid

SUMMARY:
The goal of this clinical research study is to learn if treatment with Temodar (temozolomide), Velban (vinblastine), Cisplatin, Proleukin (interleukin-2), Intron-A (interferon alpha), and thalidomide can help to control melanoma that has spread to other parts of the body. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
Some of the drugs in this study have been used with DTIC (Dacarbazine) in the past to control Melanoma that has spread to other parts of the body. However, in most of those cases, the duration of these results are limited and ineffective to control or prevent spread of the disease into the brain, the membranes that cover the brain, the spinal cord, and the nerve roots. In this study, temozolomide is being used instead of DTIC. Temodar has been proven to be one of the most effective therapeutic agents to control malignancies in the brain. Thalidomide is designed to decrease the formation of new blood vessels that feed tumors.

The treatment plan for this study is divided in two parts. The first part of this study (induction therapy) is done to try to get your disease under control. The second part of this study (maintenance therapy) is to maintain or improve the results of the first part of the treatment plan.

Induction Therapy:

Induction therapy includes three 5-day courses of treatment with thalidomide, temozolomide, vinblastine, cisplatin, interleukin-2, and interferon-alpha. The courses are repeated in cycles of three to four weeks depending on recovery from side effects from the previous course of treatment.

All of the drugs that are given through a vein will be given through a catheter (plastic tube) inserted in a vein in one of your arms or into the vein that runs underneath the collar bone and threaded into the central vein in the upper part of the chest.

You will be admitted in the hospital on Day 0. You will start receiving liquids (hydration) and be prepared to start temozolomide on day 1 of the admission. It is anticipated that you will remain in the hospital for one week. Depending on degree of side effects a longer stay in the hospital may be required.

Temozolomide will be given by mouth on the first day of the treatment every 4 hours for three doses. A fourth dose may be considered with later courses of treatment if it is well tolerated.

Vinblastine will be given through the catheter on Days 1,2,3 and 4 of the cycle. The infusion should last between 15 to 30 minutes.

Cisplatin will be given through the catheter on Days 1,2,3 and 4 of the cycle. The infusion should last between 45 to 120 minutes. Care will be given to fully hydrate the body to decrease chances for kidney damage.

Thalidomide will be given by mouth once a day throughout the cycle of treatment. It is given as a single dose starting on Day 0, the day before the start of the temozolomide, and then every day for the entire cycle.

Interleukin-2 will be given as continuous infusion through the catheter over 24 hours for four days in a row (over 96 hours). It will be given from Day 1 through Day 5 of the cycle.

Interferon alpha will be given as "an insulin-type injection" under the skin, into the fatty tissue, once a day on Days 1,2,3,4 and 5 of each cycle

You will receive up to 3 courses of induction therapy. The courses will be repeated in cycles of 3-4 weeks depending on adequate recovery from the side effects. If you have stable disease or improved disease, you will go on to receive maintenance therapy.

Maintenance Therapy:

Long-term daily treatment with the study drugs will be given for six 4-week cycles.

Temozolomide will be given by mouth daily for 21 days (3 weeks). This will be followed by one week without Temozolomide treatment. This makes up one cycle of treatment.

Interleukin-2 and interferon alpha will be given during the one week of rest from temozolomide. This will require one week of hospitalization. Interleukin-2 is given as a continuous infusion through the catheter over the first 5 days. The first day the dose will be high and it will be decreased slowly to a lower dose on the last 3 days. The interferon alpha will be given as an injection in the fatty tissues under the skin once a day for 5 days on the same days the interleukin-2 is given.

Thalidomide will be given by mouth once a day every day for the full 4-week cycle.

Supportive care with medications for fever, chills, nausea, vomiting, diarrhea, will be given during treatment. You will also be given fluids with appropriate electrolytes to replenish blood levels and to replenish blood volume to help the kidneys.

How you respond to treatment will be evaluated with computed tomography (CT) scans and magnetic resonance images (MRIs) of the brain. This will occur after the second course and third course of induction therapy and then after the third and sixth courses of maintenance therapy and periodically until off study.

You will be requested to complete a questionnaire to evaluate your quality of life before treatment starts, at the end of Cycles 2 and 3 of induction therapy, and at the end of Cycles 3 and 6 of maintenance therapy.

You will be taken off study if the disease gets worse or intolerable side effects occur. Should you be taken off study early, a long term follow-up will be requested.

For those patients who complete the treatment, radiographic evaluation with body CT scans and brain MRI will be done. They will have physical exams, and blood tests (1 to 2 tablespoons per visit) every 3 months for the first year, every 4 months for the second year, every 6 months up to the 5th year, and then once a year.

A total of 60 patients will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically documented diagnosis of advanced stage IV or unresectable stage III melanoma are eligible.
2. They should have recurrent melanoma with measureable or evaluable sites of disease in order to assess the response to treatment by Response Evaluation Criteria In Solid Tumors (RECIST) criteria.
3. Patients between 18 years of age and 65 years of age with an expected survival greater than 8 weeks and a Karnofsky performance status of 50% or better or an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 will be eligible.
4. They should have normal blood counts with a white blood count (WBC) count of more than or equal to 3000/mm^3 an absolute neutrophil count of more than or equal to 1500/mm^3 and a platelet count of more than 100,000/mm^3 and have no impairment of renal function (serum creatinine of less than 1.6 mg/dl), hepatic function (serum bilirubin level of < 1.2 mg/dl) and no evidence of significant cardiac or pulmonary dysfunction.
5. They should have no significant intercurrent illness such as an active infection, uncontrolled psychiatric illness, hypercalcemia (calcium > 11 mg), or active GI bleeding.
6. They should not have been exposed to any previous chemotherapy or isolation perfusion for malignant melanoma and have had no previous exposure to interleukin-2. Prior adjuvant interferon is permitted. Prior radiation therapy for metastatic melanoma is permitted provided the patient has un-irradiated metastatic sites for response evaluation and has fully recovered from its toxicity.

Exclusion Criteria:

1. Patients with brain and/or bone metastases only.
2. Patients with symptomatic central nervous system involvement by melanoma either as brain metastasis by MRI or spinal cord compression. Patients with brain metastases are not eligible unless their disease can be resected, it is asymptomatic, not associated with cerebral edema, or they are clinically stable after radiation and off corticosteroid therapy for 4 weeks. No major surgery or RT within 21 days before starting of treatment.
3. Patients with significant cardiac illness such as symptomatic coronary artery disease or previous history of myocardial infarction, impaired left ventricle function (EF <55%) on account of any organic disease such as hypertension or valvular heart disease or serious cardiac arrhythmia requiring therapy. Patients with an electrocardiogram (EKG) disclosing an absolute QT interval >460 msec in the presence of serum potassium >/=4.0 mEq/L and magnesium >/= 1.8 mg/dL. Patients with heart rate less than 50.
4. Patients with significant impairment of pulmonary function on account of chronic bronchitis or chronic obstructive pulmonary disease (COPD) which has resulted in impairment of vital capacity of Left Ventricular Ejection Fraction (FE VI) to <75% of predicted normal values.
5. Patients with symptomatic effusions on account of pleural, pericardial or peritoneal metastases of melanoma.
6. Patients who are unable to stay in Houston to receive therapy (first cycle) and be able to return for follow-up visits as required by this study.
7. Patients with a history of second malignant tumor, other than the common skin cancers - basal and squamous carcinomas, within the past 5 years and uncertainty about the histological nature of the metastatic lesions.
8. Patients with history of deep vein thrombi (DVT) or pulmonary embolism (PE) are excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas E. Papadopoulos, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 14, 2007 through July 9, 2009. All participants recruited at UT MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Biochemotherapy With Temozolomide
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Biochemotherapy With Temozolomide
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 43 [35 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP)
Description: TTP defined as the time from date of first dose of study medication to first documentation of objective tumor progression in days. Response evaluation by Response Evaluation Criteria in Solid Tumors (RECIST) done following 2 cycles and 3 cycles. Progression is defined, using RECIST, as a measurable increase in the smallest dimension of any target or non-target lesion, or the appearance of new lesions, since baseline.
Time Frame: Following two 21 day cycles until disease progression
Measure: Geometric Mean (Full Range); unit: days
Arm/Group | Biochemotherapy With Temozolomide
Number analyzed (Participants) | 5
days | 93.2 [44 to 164]

2. Secondary Outcome: Number of Participants With Response
Description: Response evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: Following each 21 day cycles
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year and 7 months
Arm/Group | Biochemotherapy With Temozolomide
Serious Adverse Events (participants affected / at risk) | 5/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biochemotherapy With Temozolomide (N=5)
Fatigue (General disorders) | 4
Fever/rigor (Infections and infestations) | 1
Neutropenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Hemoglobin Level (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Biochemotherapy With Temozolomide (N=5)
Fatigue (General disorders) | 5
Anorexia (Gastrointestinal disorders) | 4
Fever/rigor (Infections and infestations) | 5
Hypotension (Blood and lymphatic system disorders) | 4
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 4
Skin Rash (Skin and subcutaneous tissue disorders) | 3
Peripheral Neuropathy (Nervous system disorders) | 1
Fluid retention (Vascular disorders) | 5
Renal dysfunction (Creatinine) (Renal and urinary disorders) | 3
Hypomagnesemia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Hemoglobin Level (Blood and lymphatic system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No